CLINICAL TRIAL: NCT05711901
Title: Multicenter Observational Prospective Study of the Efficacy and Safety of Selective Lipopolysaccharide Hemosorption Using the Efferon LPS Device in Maternal Sepsis Complicated by Organ Dysfunction and/or Septic Shock
Brief Title: Selective Lipopolysaccharide Hemosorption in Maternal Sepsis
Acronym: MINERVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2022-01
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Maternal sepsIs
Keywords: septic shock; maternal sepsIs; lipopolysaccharide sorption; obstetric sepsis
MeSH Terms: conditions — Pregnancy Complications, Infectious; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Multicenter prospective study with a control group to evaluate the efficacy and safety of LPS sorption using the Efferon LPS device in postpartum sepsis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Baseline therapy (No Intervention): Basic therapy - the routine practice of an institution for the treatment of patients with maternal sepsis
- Experimental: Basic therapy + Efferon LPS (Experimental): Basic therapy is a routine practice of the institution for the treatment of patients with maternal sepsis plus extracorporeal hemoperfusion therapy (Efferon LPS)
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Hemoperfusion using continuous extracorporeal LPS adsorption with Efferon LPS therapeutic device during a period of 12h immediately following admission to the intensive care unit
  Arms: Experimental: Basic therapy + Efferon LPS

SUMMARY:
One of the major health problems in the world is sepsis, the number of cases of which, according to WHO, annually reaches 20-30 million.

The prevalence and frequency of obstetric sepsis are quite pronounced. Thus, in Europe, up to 500,000 cases of sepsis are registered annually. In Russia, the frequency of obstetric purulent-inflammatory diseases in the structure of maternal mortality ranges from 5 to 26%, according to some data - up to 45-75%. In the structure of maternal mortality, this pathology is in second or third place. Numerous studies have shown that the use of extracorporeal sorption methods that eliminate endotoxin and cytokines improves the results of treatment of patients with septic shock. The main goal of the study was to obtain new data on the efficacy and safety of using the Efferon LPS device for hemosorption of lipopolysaccharides during extracorporeal detoxification in patients with obstetric sepsis.

DETAILED DESCRIPTION:
One of the major health problems in the world is sepsis, the number of cases of which, according to WHO, annually reaches 20-30 million. One third of patients admitted to the ICU were patients with infection, a fifth of whom developed septic shock, the proportion of hospital sepsis was 46.6%, and death occurred in 30.4% of patients with infection.

The prevalence and incidence of obstetric sepsis is also pronounced. In Europe, up to 500,000 cases of sepsis are registered annually. In Russia, the frequency of obstetric purulent-inflammatory diseases in the structure of maternal mortality ranges from 5 to 26%, according to some data - up to 75%. In the structure of maternal mortality, this pathology is in second or third place.

Most often, postpartum sepsis occurs against the background of endometritis (90%), much less often against the background of a wound infection, mastitis, urinary tract infection (apostematous nephritis) or post-injection abscess. Every year, one million newborns die due to maternal infections, in particular maternal sepsis. Endotoxin, one of the most potent mediators of sepsis, is found in high concentrations in about 50% of patients with septic shock.

Despite clear progress in intensive care, the prognosis in patients with endotoxemia and septic shock remains unfavorable.

Hemoperfusion or hemoadsorption is a method of extracorporeal removal of toxic substances from the blood by their adsorption on a porous material. The hemosorption method can be a good addition or replacement to the classical methods of hemofiltration and hemodialysis, if the diffusion or convection of toxic substances through the membrane is not effective enough. Currently, using hemosorbents based on highly cross-linked copolymers of styrene and divinylbenzene, it is possible to remove endo- and exotoxins in acute and chronic renal and hepatic insufficiency, eliminate intoxication with pharmacological drugs, drugs and poisons, and also remove cytokines that are formed in excess during sepsis and systemic inflammatory diseases. syndrome of another etiology.

Numerous studies have shown that the use of endotoxin-eliminating methods of extracorporeal sorption improves outcomes in patients with sepsis and septic shock.

Efferon LPS is a device for extracorporeal blood purification by direct hemoperfusion. Detoxification is carried out by selective sorption of lipopolysaccharides (bacterial endotoxins).

The purpose of this observational study is to evaluate the efficacy and safety of multimodal (lipopolysaccharide + cytokine) sorption using the Efferon LPS device in patients with obstetric sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* An established diagnosis of sepsis according to the criteria for SEPSIS-3, most likely Gram-negative etiology, at the time of inclusion.
* No more than 12 hours from the time of setting DS - Sepsis and/or Septic Shock.

In case of septic shock:

• Hypotension requiring vasopressor support for at least 2 hours continuously and no more than 12 hours.

In the absence of Septic shock, but in the presence of suspicion of sepsis (before the detection of flora) and organ dysfunction, inclusion in the clinical trial is based on 2 of the 4 SIRS criteria,

• SOFA ≥ 4 points.

Exclusion Criteria:

* Inability to obtain informed consent from the patient, family member or legal representative,
* The presence of a focus of non-sanitized surgical infection,
* The use of other methods of extracorporeal removal of LPS and inflammatory mediators in the treatment of septic shock (hemofilters with highly permeable and surface-modified membranes)
* In Septic Shock, failure to achieve or maintain a minimum mean arterial pressure (MAP) ≥ 65 mmHg. Art., despite vasopressor therapy and infusion therapy for 24 hours,
* End-stage renal disease and need for chronic dialysis.
* Acute pulmonary embolism
* Transfusion reaction,
* Severe congestive heart failure,
* Uncontrolled bleeding (acute blood loss in the last 24 hours),
* Severe granulocytopenia (white blood cell count less than 500 cells/mm3),
* Any other condition that, in the opinion of the investigator, would prevent the patient from being a suitable candidate for inclusion in the study (eg terminal chronic disease).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon LPS hemoperfusion on SOFA (Sequential Organ Failure Assessment) scores in patients with obstetric sepsis. | 1-72 hours
  The value of indicators on the SOFA (Sequential Organ Failure Assessment) scale every 24 hours ± 1 hour from the start of hemoperfusion (0 hour) to 72 hours. The SOFA index is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall index, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. With a score of no more than 12, multiple organ dysfunctions are assumed, 13-17 points indicate the transition of dysfunction to insufficiency, a score of about 24 indicates a high probability of death. The lower the SOFA index, the less pronounced organ failure and the better the patient's survival prognosis.
The effect of Efferon-LPS hemoperfusion on hemodynamic parameters in patients with obstetric sepsis | Time (number of hours) from enrollment in the study to the end of vasopressor support during 14 days of follow-up
  Event criteria: end of vasopressor support (maintenance of effect for 4 hours)

SECONDARY OUTCOMES:
Effect of LPS Efferon hemoperfusion on endotoxin activity | 1-72 hours
  Value of endotoxin levels every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours
Effect of the Efferon LPS hemoperfusion on pulmonary oxygen metabolism function | 1-72 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours.
Effect of the Efferon LPS hemoperfusion on the length of stay in the ICU | 1-14 days
  Time (number of days) from enrollment in the study to transfer from the ICU within 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Pyregov, PhD, MD, Principal Investigator — Moscow Regional Perinatal Center
Locations (7):
- Russia (7):
  - Krasnoyarsk Regional Clinical Hospital, Krasnoyarsk
  - Moscow Regional Perinatal Center, Moscow
  - National Medical Research Center named after V.I. Kulakov, Moscow
  - Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod
  - Perm regional clinical hospital, Perm
  - Surgut District Clinical Center for Maternity and Childhood Health, Surgut
  - Perinatal Center of the Tyumen Region, Tyumen